CLINICAL TRIAL: NCT05119270
Title: Comparison of Corneal Endothelial Cell Loss and Cumulative Dissipated Energy Between Femtosecond Laser Assisted Cataract Surgery and Standard Phacoemulsification With the Active Sentry or OZil Handpiece
Brief Title: Comparison of Phacoemulsification and Corneal Damage Between FLACS and Standard Phaco With Two Handpieces
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 21.225
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Corneal Endothelial Cell Loss; Cataract; Astigmatism
Keywords: Corneal Endothelial Cell Loss; Centurion Vision System; Infiniti Vision System; cumulative dissipated energy; Phacoemulsification; Active Sentry handpiece; Laser Therapy; Ozil handpiece
MeSH Terms: conditions — Corneal Endothelial Cell Loss; Cataract; Astigmatism

STUDY DESIGN:
Intervention Model Description: 3 groups will be compared:
  * Group 1: 30 participants suffering from cataract who are candidates for femtosecond laser assisted cataract surgery
  * Group 2: 30 participants suffering from cataract who are candidates for traditional cataract surgery with the Active Sentry handpiece
  * Group 3: 30 participants suffering from cataract who are candidates for traditional cataract surgery with the OZil handpiece
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Femtosecond laser assisted cataract surgery with Active Sentry handpiece (Experimental): Participants suffering from cataract who are candidates for femtosecond laser assisted cataract surgery
  Interventions: Device: Femtosecond laser assisted cataract surgery with Active Sentry handpiece
- Standard phacoemulsification with the Active Sentry handpiece (Experimental): Participants suffering from cataract who are candidates for standard phacoemulsification with the new Active Sentry handpiece
  Interventions: Procedure: Standard phacoemulsification with the Active Sentry handpiece
- Standard phacoemulsification with the OZil handpiece (Experimental): Participants suffering from cataract who are candidates for standard phacoemulsification with the traditional OZil handpiece
  Interventions: Procedure: Standard phacoemulsification with the OZil handpiece

INTERVENTIONS:
Device: Femtosecond laser assisted cataract surgery with Active Sentry handpiece — The LenSx laser (Alcon Laboratories Inc., USA) automates key steps in the procedure including capsulorhexis, incision making and phaco. The Frequency Domain - Optical Coherence Tomography (FD-OCT) optical imaging system provides high-resolution, real-time visualization of ocular structures and their dimensions. The device sends the results to the interface which programs the laser and indicates the exact location, size and depth of the desired incisions.
  Diagnostic tests:
  1. Corneal topography: OPD-Scan Corneal topography photography, taken by specular reflection (OPD-Scan) by measuring corneal curvature, thickness and topography
  2. Pachymetry: precise measurement of the thickness of the cornea using a pachymeter
  3. Specular microscopy : Qualitative and quantitative analysis of the corneal endothelium.
  Arms: Femtosecond laser assisted cataract surgery with Active Sentry handpiece
Procedure: Standard phacoemulsification with the Active Sentry handpiece — Phacoemulsification is done by using the Active Sentry handpiece to allow for a better control of the intraocular pressure throughout the surgery.
  Diagnostic tests:
  1. Corneal topography: OPD-Scan Corneal topography photography, taken by specular reflection (OPD-Scan) by measuring corneal curvature, thickness and topography
  2. Pachymetry: precise measurement of the thickness of the cornea using a pachymeter
  3. Specular microscopy : Qualitative and quantitative analysis of the corneal endothelium.
  Arms: Standard phacoemulsification with the Active Sentry handpiece
Procedure: Standard phacoemulsification with the OZil handpiece — Phacoemulsification is done by using the traditional OZil handpiece that allows rotational movement of the phaco tip.
  Diagnostic tests:
  1. Corneal topography: OPD-Scan Corneal topography photography, taken by specular reflection (OPD-Scan) by measuring corneal curvature, thickness and topography
  2. Pachymetry: precise measurement of the thickness of the cornea using a pachymeter
  3. Specular microscopy : Qualitative and quantitative analysis of the corneal endothelium.
  Arms: Standard phacoemulsification with the OZil handpiece

SUMMARY:
The main goal of this study is to compare traditional cataract surgery with two new technologies: the femtosecond laser and the new Active Sentry handpiece.

The femtosecond laser is used in several fields of ophthalmology and allows to automate multiple key steps of cataract surgery.

The new generation of handpiece called Active Sentry has the particularity to detect the pressure inside the eye in real time and to adjust it to avoid large variations.

Theses technologies would potentially increase the efficacy and safety of standard cataract surgery. This study therefore aims at evaluating the differences in cumulative dissipated energy and endothelial cell loss between femtosecond laser assisted cataract surgery with the new Active Sentry handpiece compared to standard phaco with new (Active Sentry) or older handpieces (OZil).

DETAILED DESCRIPTION:
Phacoemulsification (phaco) has been the standard technique for cataract surgery for several decades. It involves the removal of the lens nucleus after ultrasound fragmentation. Recently, Femtosecond Laser Assisted Cataract Surgery (FLACS) has become a new popular method amongst ophthalmologists.

The femtosecond laser (LFS) is a new technology that is being used for cataract surgery. The LFS has a femtosecond pulse duration, which reduces damage to collateral tissue and increases the efficacy and safety of the procedure. The LenSx laser (Alcon Laboratories Inc., USA) is one of the most widely used LFS for cataract surgery and is part of the CENTURION Vision system. The LFS automates key steps in the procedure including capsulorhexis, incision making and phaco, limiting human variability and potentially improving the efficiency and safety of the surgery. The Frequency Domain - Optical Coherence Tomography (FD-OCT) optical imaging system provides high-resolution, real-time visualization of ocular structures and their dimensions. The device sends the results to the interface which programs the laser and indicates the exact location, size and depth of the desired incisions.

Several handpieces are used to perform phacoemulsification. The traditional handpiece is named OZil and is part of the Infiniti Vision System (Alcon Laboratories Inc.) which was introduced in 2006 and has since revolutionized the phaco technique with its new rotational technology. This handpiece increased phaco efficacy by reducing core fragment repulsion, collateral tissue damage, and the amount of energy required. However, a new generation of handpiece called Active Sentry (Alcon Inc.), which is part of the new Active Fluidics technology, has now the added feature of detecting the pressure inside the eye in real time and adjusting it to avoid significant variations. This handpiece can also decrease the amount of fluid and energy used during the procedure, increasing the efficacy and safety of phacoemulsification.

Different methods to quantify the collateral damage caused by cataract surgeries are the count of endothelial cell loss (ECL) as well as the amount of energy required to fragment the lens (CDE: cumulative dissipated energy). FLACS may reduce the CDE required during phaco, thereby reducing the damage to the cornea of the eye (including the loss of endothelial cells of the cornea).

Despite a large number of publications on this topic, recent meta-analyses on the effect of FLACS on ECL and CDE were found to be inconsistent. Few studies have demonstrated a decrease in ECL as well as CDE required in patients undergoing FLACS when compared to standard phaco, but long-term results were not conclusive.

Given the novelty of the Active Sentry handpiece, little data on this new device exists in the literature. Based on what was found in the literature, this study will be the first to compare the following techniques: FLACS with Active Sentry, traditional phaco with Active Sentry, and traditional phaco with OZil.

The investigators hypothesize that the new FLACS technique will reduce the CDE required during phacoemulsification, thereby reducing the damage caused the cornea (i.e. loss of endothelial corneal cells).

In addition, the investigators hypothesize that patients undergoing standard phacoemulsification with the Active Sentry handpiece will have less corneal endothelial cell damage and require less CDE than participants undergoing standard phacoemulsification with OZil.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (over 18 years of age)
* Patients undergoing uncomplicated cataract surgery with intraocular lens implantation
* Ability to provide informed consent;
* Ability to be followed for the entire duration of the study.

Exclusion Criteria:

* Minor patient (under 18 years of age)
* Unable to give informed consent
* Unable to be followed for the duration of the study
* Another surgery combined with cataract extraction
* History of ocular surgery
* Patient with concomitant ocular diseases other than cataract (such as corneal, retinal, or glaucoma diseases)
* Irregular corneal astigmatism or keratoconus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Corneal endothelial cell loss (Specular microscopy) | Baseline, 1 month, 3 months
  Change in corneal endothelial cells count after cataract surgery
Cumulative dissipated energy | Peroperatively
  Amount of energy used during phacoemulsification

SECONDARY OUTCOMES:
Central corneal thickness | Baseline, 1 month, 3 months
  Change in central thickness of the corneal measured by a pachymeter.
Postoperative residual astigmatism | Baseline, 3 months
  Change in simulated keratometric values obtained by OPD-Scan.
Binocular uncorrected visual acuities for distance (6 meters) | Baseline, 1 day, 2 weeks, 1 month, 3 months
  Evaluation of visual acuity change, measured using the Snellen chart.
Patient reported visual disturbances | Baseline, 3 months
  Evaluation of patient reported visual disturbances using a validated questionnaire for visual disturbances (CaT-PROM5)

CONTACTS AND LOCATIONS:
Overall Officials: Georges Durr, MD, FRCSC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelman CD. Phaco-emulsification and aspiration. A new technique of cataract removal. A preliminary report. Am J Ophthalmol. 1967 Jul;64(1):23-35. No abstract available. PMID 6028631
- [Background] Nagy Z, Takacs A, Filkorn T, Sarayba M. Initial clinical evaluation of an intraocular femtosecond laser in cataract surgery. J Refract Surg. 2009 Dec;25(12):1053-60. doi: 10.3928/1081597X-20091117-04. PMID 20000286
- [Background] Bille JF, editor. High Resolution Imaging in Microscopy and Ophthalmology: New Frontiers in Biomedical Optics [Internet]. Cham (CH): Springer; 2019. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK554051/ PMID 32091677
- [Background] Liu Y, Zeng M, Liu X, Luo L, Yuan Z, Xia Y, Zeng Y. Torsional mode versus conventional ultrasound mode phacoemulsification: randomized comparative clinical study. J Cataract Refract Surg. 2007 Feb;33(2):287-92. doi: 10.1016/j.jcrs.2006.10.044. PMID 17276271
- [Background] Solomon KD, Lorente R, Fanney D, Cionni RJ. Clinical study using a new phacoemulsification system with surgical intraocular pressure control. J Cataract Refract Surg. 2016 Apr;42(4):542-9. doi: 10.1016/j.jcrs.2016.01.037. PMID 27113876
- [Background] Al-Mohtaseb Z, He X, Yesilirmak N, Waren D, Donaldson KE. Comparison of Corneal Endothelial Cell Loss Between Two Femtosecond Laser Platforms and Standard Phacoemulsification. J Refract Surg. 2017 Oct 1;33(10):708-712. doi: 10.3928/1081597X-20170731-01. PMID 28991340
- [Background] Chen X, Xiao W, Ye S, Chen W, Liu Y. Efficacy and safety of femtosecond laser-assisted cataract surgery versus conventional phacoemulsification for cataract: a meta-analysis of randomized controlled trials. Sci Rep. 2015 Aug 13;5:13123. doi: 10.1038/srep13123. PMID 26269445
- [Background] Ye Z, Li Z, He S. A Meta-Analysis Comparing Postoperative Complications and Outcomes of Femtosecond Laser-Assisted Cataract Surgery versus Conventional Phacoemulsification for Cataract. J Ophthalmol. 2017;2017:3849152. doi: 10.1155/2017/3849152. Epub 2017 Apr 30. PMID 28540082
- [Background] Saeedi OJ, Chang LY, Ong SR, Karim SA, Abraham DS, Rosenthal GL, Hammer A, Spagnolo BV, Betancourt AE. Comparison of cumulative dispersed energy (CDE) in femtosecond laser-assisted cataract surgery (FLACS) and conventional phacoemulsification. Int Ophthalmol. 2019 Aug;39(8):1761-1766. doi: 10.1007/s10792-018-0996-x. Epub 2018 Jul 27. PMID 30054849
- [Background] Bascaran L, Alberdi T, Martinez-Soroa I, Sarasqueta C, Mendicute J. Differences in energy and corneal endothelium between femtosecond laser-assisted and conventional cataract surgeries: prospective, intraindividual, randomized controlled trial. Int J Ophthalmol. 2018 Aug 18;11(8):1308-1316. doi: 10.18240/ijo.2018.08.10. eCollection 2018. PMID 30140634
- [Background] Krarup T, Holm LM, la Cour M, Kjaerbo H. Endothelial cell loss and refractive predictability in femtosecond laser-assisted cataract surgery compared with conventional cataract surgery. Acta Ophthalmol. 2014 Nov;92(7):617-22. doi: 10.1111/aos.12406. Epub 2014 Jun 2. PMID 24888390
- [Background] Jiraskova N, Stepanov A. OUR EXPERIENCE WITH ACTIVE SENTRY AND CENTURION OZIL HANDPIECES. Cesk Slov Oftalmol. 2021 Winter;77(1):18-21. doi: 10.31348/2021/1. PMID 33740863
- [Background] Ho JW, Afshari NA. Advances in cataract surgery: preserving the corneal endothelium. Curr Opin Ophthalmol. 2015 Jan;26(1):22-7. doi: 10.1097/ICU.0000000000000121. PMID 25415300